CLINICAL TRIAL: NCT04914299
Title: Positive Intelligence - Prospective Study Evaluating a Novel Mobile App Based Preventive Behavioral Intervention for Perinatal Mood Disorders
Brief Title: Prospective Study Evaluating a Novel Mobile App Based Preventive Behavioral Intervention for Perinatal Mood Disorders
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Positive Intelligence Inc. (Unknown)
Responsible Party: Principal Investigator, Shay Erisson, Physician, Obstetrics and Gynecology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021P001387
Record Dates: First submitted 2021-05-31; First posted 2021-06-04 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Perinatal Depression; Perinatal Anxiety
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Two groups: One receives a novel mobile-App based intervention and the other groups receives standard of care (psychoeducation about postpartum depression, referral and monitoring).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A novel mobile-App based intervention (Experimental): An App-based "positive intelligence" intervention consisting of 6 weeks of weekly videos and support group sessions, and 6 weeks of daily App-guided practices.
  Interventions: Behavioral: App-based "positive intelligence" intervention; Behavioral: Standard of care
- Standard of Care (Active Comparator): Standard prenatal care and follow up
  Interventions: Behavioral: Standard of care

INTERVENTIONS:
Behavioral: App-based "positive intelligence" intervention — A 6 weeks App-guided and support-group based "positive intelligence" cognitive behavioral intervention in addition to standard prenatal and postnatal care
  Arms: A novel mobile-App based intervention
Behavioral: Standard of care — Standard prenatal and postnatal care(Providing psychoeducation and referral to psychotherapy or pharmacotherapy based on participant's symptoms).

SUMMARY:
The primary aim of the study is to investigate whether a novel mobile App-based behavioral intervention in pregnant women can: (1) prevent and/or decrease the incidence of perinatal mood disorders (2) decrease the severity and/or duration of perinatal mood disorders in affected participants (3) increase access of pregnant women to behavioral intervention and support tools (4) increase the satisfaction of pregnant women with their prenatal care.

DETAILED DESCRIPTION:
Perinatal depression is an episode of major or minor depression that occurs during pregnancy or in the 12 months after birth; it affects about 10% of new mothers. Postpartum depression accounts for 12.5% of psychologically related hospitalizations among women.

In 2019, the United States Preventive Services Task Force (USPSTF) recommended screening pregnant women to identify those at risk for perinatal depression and refer them for counseling. The USPSTF recommendation is based on growing literature indicating that counseling women at risk for perinatal depression reduce the risk of having an episode of major depression by 40%.

Supporting that, multiple studies have shown that cognitive-behavioral intervention and mental health care adjuvant therapy can effectively improve the condition of patients with postpartum depression. Finally, access to care has also been shown to be an important factor in determining the success of any intervention. Women across high and low-risk groups often have barriers to treatment due to stigma, shame, and fear to disclose symptoms to health providers

In this research, the investigators aim to investigate whether a novel mobile App-based behavioral intervention can meaningfully increase access and demonstrate a beneficial effect in preventing anxiety and depression in the postpartum period. Furthermore and adding to the existing literature in post-partum depression, this study aims to investigate the role of "positive intelligence", an integrative positive cognitive behavioral therapy, as a tool in the prevention and treatment of perinatal mood disorders.

ELIGIBILITY:
Inclusion Criteria:

* Able to read and speak English
* Have a low-risk singleton pregnancy with more than 24 weeks of gestation
* Have smartphone with internet access
* Failure to meet criteria for a diagnosis of MDD in the last two months

Exclusion Criteria:

* Physical or mental disorders which would interfere with their ability to participate in the study
* High-risk pregnancy
* Give birth to a newborn at still-birth or a newborn with congenital anomalies and/or Medical complications that require special care in hospital
* Infant has a birth weight lower than 2,500 grams
* Infant has a 5-minute Apgar score lower than 7

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Postpartum Depression Symptoms | 3rd trimester pregnancy till 6 months postpartum
  Postpartum Depression Symptoms measured by Edinburgh Postnatal Depression Scale postpartum. Scale 1-30,with 0 indicating no symptoms, and 30 indicating the highest severity of symptoms.

SECONDARY OUTCOMES:
Completion of App-based intervention program | 6 weeks postpartum
  Self reported completion of App based 6 weeks training program.
Patient Satisfaction | 6 weeks postpartum to 6 months postpartum
  Patient satisfaction measured by Client Satisfaction Questionnaire scale. scale 8-32, with higher scores indicate greater satisfaction.
Generalized Anxiety Symptoms | 3rd trimester pregnancy till 6 months postpartum
  Anxiety Symptoms measured by Generalized Anxiety Scale. scale 0-21, with with 0 indicating no symptoms, and 21 indicating the highest severity of symptoms.
Patient depression symptoms and severity | 3rd trimester pregnancy till 6 months postpartum
  Depression Symptoms measured by Patient Health Questionnaire scale. Scale 0-27, with 0 indicating no symptoms, and 27 indicating the highest severity of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Shay Erisson, MD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] The American College of Obstetricians and Gynecologists Committee Opinion no. 630. Screening for perinatal depression. Obstet Gynecol. 2015 May;125(5):1268-1271. doi: 10.1097/01.AOG.0000465192.34779.dc. PMID 25932866
- [Background] ACOG Committee Opinion No. 757: Screening for Perinatal Depression. Obstet Gynecol. 2018 Nov;132(5):e208-e212. doi: 10.1097/AOG.0000000000002927. PMID 30629567
- [Background] ACOG Committee Opinion No. 736: Optimizing Postpartum Care. Obstet Gynecol. 2018 May;131(5):e140-e150. doi: 10.1097/AOG.0000000000002633. PMID 29683911
- [Background] Morrell CJ, Sutcliffe P, Booth A, Stevens J, Scope A, Stevenson M, Harvey R, Bessey A, Cantrell A, Dennis CL, Ren S, Ragonesi M, Barkham M, Churchill D, Henshaw C, Newstead J, Slade P, Spiby H, Stewart-Brown S. A systematic review, evidence synthesis and meta-analysis of quantitative and qualitative studies evaluating the clinical effectiveness, the cost-effectiveness, safety and acceptability of interventions to prevent postnatal depression. Health Technol Assess. 2016 May;20(37):1-414. doi: 10.3310/hta20370. PMID 27184772
- [Background] US Preventive Services Task Force; Curry SJ, Krist AH, Owens DK, Barry MJ, Caughey AB, Davidson KW, Doubeni CA, Epling JW Jr, Grossman DC, Kemper AR, Kubik M, Landefeld CS, Mangione CM, Silverstein M, Simon MA, Tseng CW, Wong JB. Interventions to Prevent Perinatal Depression: US Preventive Services Task Force Recommendation Statement. JAMA. 2019 Feb 12;321(6):580-587. doi: 10.1001/jama.2019.0007. PMID 30747971
- [Background] Zlotnick C, Johnson SL, Miller IW, Pearlstein T, Howard M. Postpartum depression in women receiving public assistance: pilot study of an interpersonal-therapy-oriented group intervention. Am J Psychiatry. 2001 Apr;158(4):638-40. doi: 10.1176/appi.ajp.158.4.638. PMID 11282702
- [Background] Zlotnick C, Miller IW, Pearlstein T, Howard M, Sweeney P. A preventive intervention for pregnant women on public assistance at risk for postpartum depression. Am J Psychiatry. 2006 Aug;163(8):1443-5. doi: 10.1176/ajp.2006.163.8.1443. PMID 16877662
- [Background] McFarlane E, Burrell L, Duggan A, Tandon D. Outcomes of a Randomized Trial of a Cognitive Behavioral Enhancement to Address Maternal Distress in Home Visited Mothers. Matern Child Health J. 2017 Mar;21(3):475-484. doi: 10.1007/s10995-016-2125-7. PMID 27535131
- [Background] Pessagno RA, Hunker D. Using short-term group psychotherapy as an evidence-based intervention for first-time mothers at risk for postpartum depression. Perspect Psychiatr Care. 2013 Jul;49(3):202-9. doi: 10.1111/j.1744-6163.2012.00350.x. Epub 2012 Aug 17. PMID 23819670
- [Background] O'Connor E, Senger CA, Henninger ML, Coppola E, Gaynes BN. Interventions to Prevent Perinatal Depression: Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2019 Feb 12;321(6):588-601. doi: 10.1001/jama.2018.20865. PMID 30747970
- [Background] Liu H, Yang Y. Effects of a psychological nursing intervention on prevention of anxiety and depression in the postpartum period: a randomized controlled trial. Ann Gen Psychiatry. 2021 Jan 4;20(1):2. doi: 10.1186/s12991-020-00320-4. PMID 33397393
- [Background] Avalos LA, Raine-Bennett T, Chen H, Adams AS, Flanagan T. Improved Perinatal Depression Screening, Treatment, and Outcomes With a Universal Obstetric Program. Obstet Gynecol. 2016 May;127(5):917-925. doi: 10.1097/AOG.0000000000001403. PMID 27054938
- [Background] Byatt N, Simas TA, Lundquist RS, Johnson JV, Ziedonis DM. Strategies for improving perinatal depression treatment in North American outpatient obstetric settings. J Psychosom Obstet Gynaecol. 2012 Dec;33(4):143-61. doi: 10.3109/0167482X.2012.728649. PMID 23194018
- [Background] Sockol LE. A systematic review and meta-analysis of interpersonal psychotherapy for perinatal women. J Affect Disord. 2018 May;232:316-328. doi: 10.1016/j.jad.2018.01.018. Epub 2018 Feb 1. PMID 29501991
- [Background] Sockol LE. A systematic review of the efficacy of cognitive behavioral therapy for treating and preventing perinatal depression. J Affect Disord. 2015 May 15;177:7-21. doi: 10.1016/j.jad.2015.01.052. Epub 2015 Feb 2. PMID 25743368
- [Background] Haga SM, Drozd F, Lisoy C, Wentzel-Larsen T, Slinning K. Mamma Mia - A randomized controlled trial of an internet-based intervention for perinatal depression. Psychol Med. 2019 Aug;49(11):1850-1858. doi: 10.1017/S0033291718002544. Epub 2018 Sep 7. PMID 30191779
- [Background] Shorey S, Ng YPM, Ng ED, Siew AL, Morelius E, Yoong J, Gandhi M. Effectiveness of a Technology-Based Supportive Educational Parenting Program on Parental Outcomes (Part 1): Randomized Controlled Trial. J Med Internet Res. 2019 Feb 13;21(2):e10816. doi: 10.2196/10816. PMID 30758289
- [Background] Goodman JH. Women's attitudes, preferences, and perceived barriers to treatment for perinatal depression. Birth. 2009 Mar;36(1):60-9. doi: 10.1111/j.1523-536X.2008.00296.x. PMID 19278385
- [Background] Smith-Nielsen J, Matthey S, Lange T, Vaever MS. Validation of the Edinburgh Postnatal Depression Scale against both DSM-5 and ICD-10 diagnostic criteria for depression. BMC Psychiatry. 2018 Dec 20;18(1):393. doi: 10.1186/s12888-018-1965-7. PMID 30572867